CLINICAL TRIAL: NCT01991444
Title: Registry Study to Evaluate the Predictive Value of a Comprehensive Geriatric Assessment With Regard to the Outcome of a Transcatheter Aortic Valve Implantation.
Brief Title: CGA-TAVI Registry to Evaluate the Predictive Value of a CGA in Predicting TAVI Outcomes
Acronym: CGA-TAVI
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Other Study IDs: U1111-1149-9951; DRKS00005436 (Other: Deutsches Register für Klinische Studien)
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TAVI patients of > 79 years: All patients undergoing transcatheter valve implantation with commercially available Edwards SAPIEN XT Transcatheter Heart Valve in participating sites.
  Routine data about the intervention (transcatheter valve Implantation) will be collected. In addition, data describing the geriatric status of the patient, including a patient questionnaire evaluating his/her Quality of life will be collected.
  Interventions: Other: TAVI

INTERVENTIONS:
Other: TAVI — no Intervention planned, Observation only

SUMMARY:
Registry study to evaluate the predictive value of a comprehensive geriatric assessment with regard to the outcome of a transcatheter aortic valve Implantation.

It will be evaluated which parts of the comprehensive geriatric assessment (CGA) are best suited to predict the therapeutic success of a heart valve Implantation in elderly ( > 80 years) Patient. Possible participants are all Patient of 80 years or above for whom the implantation of a Edwards Sapien XT aortic valve is planned

DETAILED DESCRIPTION:
Transcatheter Aortic Valve Implantation Registry with Comprehensive Geriatric Assessment

ELIGIBILITY:
Inclusion Criteria:

* Scheduled TAVI using Edwards SAPIEN XT Transcatheter Heart Valve
* Compliance with the indications of the instructions for use
* Age of at least 80 years
* Written informed consent

Exclusion Criteria:

* Presence of contraindications as to the Instructions for Use
* No possibility for a follow-up

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients undergoing transcatheter valve implantation with commercially available Edwards SAPIEN XT Transcatheter Heart Valve in participating sites.
  Routine data about the invervention (transcatheter valve Implantation) will be collected. In addition, data describing the geriatric status of the patient, including a patient questionnaire evaluating his/her Quality of life will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Comprehensive geriatric assessment | Baseline and 3 months
  Demonstrate CGA changes within 3 months after TAVI
  The CGA is an array of several different assessments with regard to frailty, comorbidities, administrative data (Silver code), Quality of life etc. Every Patient will undergo a CGA at baseline and 3 months after TAVI. Data will be analyzed to determine changes in CGA results.

SECONDARY OUTCOMES:
predictive Value of CGA Tavi | baseline
  Establish predictive value of CGA (MPI, SPPB, SilverCode) in TAVI patients for all-cause hospitalization, TAVI related hospitalization, nursing home admission
Score development | after 3 months
  Development of a comprehensive score for the assessment of TAVI patient prognosis (identifying variables from the MPI, SPPB and SilverCode that account for 80% of the predictive power of the complete set)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ungar, MD, Principal Investigator — Geriatric Cardiology and Medicine - U. of Florence
Locations (3):
- CRCHUM Montréal, Montreal, Canada
- University Medical Center, Florence, Italy
- Academisch Medisch Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ungar A, Mannarino G, van der Velde N, Baan J, Thibodeau MP, Masson JB, Santoro G, van Mourik M, Jansen S, Deutsch C, Bramlage P, Kurucova J, Thoenes M, Maggi S, Schoenenberger AW. Comprehensive geriatric assessment in patients undergoing transcatheter aortic valve implantation - results from the CGA-TAVI multicentre registry. BMC Cardiovasc Disord. 2018 Jan 4;18(1):1. doi: 10.1186/s12872-017-0740-x. PMID 29301486